CLINICAL TRIAL: NCT03141125
Title: The Effect of Ethanol Extract Physalis Angulata Linn. in Scleroderma Patients With Standard Therapy to Reduce Skin Fibrosis Based on Modified Rodnan Skin Score, Reduce Inflammation, Immunological Response and Fibrosis
Brief Title: The Effect of Ethanol Extract Physalis Angulata Linn. in Scleroderma Patients With Standard Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Principal Investigator, Sumartini Dewi, MD, Master of Health, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UI-PAL/CCD-SSc.2016
Record Dates: First submitted 2016-06-20; First posted 2017-05-04 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Scleroderma
Keywords: Erythrocyte sedimentation rate; Modified Rodnan Skin Score; B-cell Activating Factor; soluble-CD40Ligand; Procollagen Type-1 N-terminal Propeptide; Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Starch

STUDY DESIGN:
Intervention Model Description: Physalis angulata Linn. ethanol extract 3 x 250 mg
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind randomized placebo controlled trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physalis angulata ethanol extract (Experimental): Physalis angulata ethanol extract was given with dosage 3 x 250 mg/day, orally, for 3 months.
  In addition, patients also received standard therapy for scleroderma.
  Interventions: Other: Physalis angulata ethanol extract
- Placebo (Placebo Comparator): Patients received standard therapy and placebo (amylum powder) for comparator at dosage 3 x 250 mg/day, orally, for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Physalis angulata ethanol extract — Ethanol extract of physalis angulate Linn with dosage of 3x250 mg/day given orally for 3 months
  Other Names: Herba Ciplukan; Ethanol extract of Physalis angulata Linn; Ethanol extract of Physalis angulata
  Arms: Physalis angulata ethanol extract
Other: Placebo — No active component at the same dosage of 3x250 mg/day given orally for 3 months
  Other Names: Amylum
  Arms: Placebo

SUMMARY:
Study about the effect of ethanol extract physalis angulate in scleroderma patients with standard therapy to reduce skin fibrosis based on modified Rodnan Skin Score, reduce inflammation, immunological response and fibrosis: A Randomized Clinical Placebo ControlledTrial with a prospective cohort study on scleroderma outpatient clinic in Cipto Mangunkusumo Hospital in Jakarta and Hasan Sadikin Hospital in Bandung, from January 2016 to July 2017

DETAILED DESCRIPTION:
Background.

Scleroderma is a systemic autoimmune disease that can not be cured, the progression of the disease still difficult to prevent and lead to increased morbidity and mortality. Disease-modifying anti-rheumatic drugs (DMARDs) as standard immunosuppressant drugs to reduce, eliminate, inhibit inflammation and fibrosis in scleroderma patient is still less effective.

Objectives.

To evaluate the effect of ethanol extract of Physalis angulate Linn to reduce skin fibrosis based on MRSS, ESR, BAFF, sCD40L, and P1NP in scleroderma patients with standard therapy

Methods.

A Randomized, Double-Blind, Placebo-Controlled Clinical Trial on scleroderma patients with standard therapy, who admitted to Cipto Mangunkusumo Hospital Jakarta and Hasan Sadikin Hospital Bandung, from January 2016 to July 2017.

Patients must be controlled every month until three months for follow up. Subjects were divided into two parallel group, one of intervention group, and one of placebo group

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the criteria of the type of limited scleroderma diagnosis / limited or diffuse type.
2. Patients who routine control in rheumatology outpatient clinics in Ciptomangunkusumo hospital Jakarta and Hasan Sadikin hospital Bandung RSHS who received standard therapy for scleroderma with a stable dose over the past 3 months.
3. The research subjects aged 15 to 60 years.
4. Subjects with modified Rodnan Skin score ≥ 5.
5. Disease duration ≥ 1 year

Exclusion Criteria:

1. Impaired liver function with cirrhosis
2. Chronic Renal dysfunction (chronic kidney disease stages 4-5). Or creatinine levels> 2 mg / dL in the last 1 month prior to randomization.
3. Other autoimmune disease/overlap syndrome.
4. Received a steroid/prednisone >10 mg/day in the last 1 month.
5. Patients who are pregnant or breastfeeding.
6. Patients with active tuberculosis and or are being treated with anti-tuberculosis medicines.
7. Severe heart disease. (Heart Disease with impaired function according to the New York Heart Association Class III or IV)
8. History of allergies to herbal Ciplukan / Physalis angulate Linn. or a history of hypersensitivity to certain drugs.
9. Hypotension (BP <90/60 mmHg)
10. Hypoglycemia (Glucose level <70 mg / dL)
11. Do not want to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Degree of skin fibrosis based on modified Rodnan Skin Score (mRSS) | 3 months of intervention
  Clinical improvement of skin fibrosis in scleroderma patients measured by modified Improvement in skin fibrosis is defined if there is a significant reduced of mRSS.

SECONDARY OUTCOMES:
Level of P1NP serum | 3 months of intervention
  Improvement is defined if there is a significant reduced of P1NP serum level
Value of ESR | 3 months of intervention
  Improvement is defined if there is a significant reduced of ESR value
Level of BAFF serum | 3 months of intervention
  Improvement is defined if there is a significant reduced of BAFF serum level
Level of sCD40L serum | 3 months of intervention
  Improvement is defined if there is a significant reduced of sCD40L serum level.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Isbagio, MD, Prof., Study Chair — Department of Internal Medicine
Locations (2):
- Indonesia (2):
  - Hasan Sadikin Hospital, Bandung, West Java
  - Ciptomangunkusumo Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No